CLINICAL TRIAL: NCT05397769
Title: Envafolimab Plus Chemoradiotherapy for Locally Advanced Nasopharyngeal Carcinoma, a Prospective, Single Armed Phase II Trial.
Brief Title: Envafolimab Plus Chemoradiotherapy for Locally Advanced NPC, a Prospective, Single Armed Phase II Trial.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Fei Han, professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2022-203-01
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Locally Advanced Nasopharyngeal Carcinoma; Envafolimab; Induction Chemotherapy; PD-L1
MeSH Terms: interventions — envafolimab; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Envafolimab group (Experimental): Envafolimab is a PD-L1 antibody by hypodermic injection. Envafolimab will be administrated with 300mg each time, every three weeks for a total of 22 cycles since the first day of induction chemotherapy.
  Interventions: Drug: Envafolimab Plus Chemoradiotherapy

INTERVENTIONS:
Drug: Envafolimab Plus Chemoradiotherapy — Envafolimab was administrated with 300mg each time, every three weeks for a total of 22 cycles since the first day of induction chemotherapy.

SUMMARY:
Patients diagnosed with locally advanced nasopharyngeal carcinoma will be recruited in this study. All the patients will get 3 cycles of GP+ Envafolimab for the induction chemotherapy. After that, the patients will receive concurrent chemoradiotherapy. Radiotherapy will be given by IMRT, under the dose of GTVnx 68-70Gy/30-33f, 5d/w,6-7w, during which, every patient would receive 2 cycles of DDP+Envafolimab as concurrent chemotherapy. Then patients would receive Envafolimab every 3 weeks for maintenance treatment for a year, until disease progression or intolerance of treatment. . We aim to evaluate the three years progression free survival of these patients by the combination of Envafolimab with curative chemoradiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* ECOG 0-1
* histologically confirmed non-keratinizing carcinoma (WHO type II or III) of nasal pharynx
* stage III-IVa （AJCC/UICC 8th ）, untreated NPC patients
* NE≥ 1.5×10E9/L, HGB ≥ 100g/L and PLT ≥100×10E9/L
* ALT≤ 1.5 upper limit of normal (ULN), AST≤ 1.5ULN and bilirubin ≤ 1.5ULN
* creatinine<1.5×ULN

Exclusion Criteria:

* recurrent or metastatic NPC patients
* histologically confirmed keratinizing carcinoma (WHO type I) of nasal pharynx
* already received radiation or chemotherapy
* pregnant or lactating women, or women of childbearing age without birth control
* HIV (+)
* had other cancers before
* used immune checkpoint inhibitor(CTLA-4、PD-1、PD-L1 etc.) before
* complications requiring long-term treatment with immunosuppressive drugs or systemic or local use of corticosteroids with immunosuppressive dose
* with immune deficiency diseases, or a history of organ transplantation (including but not limited to: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, nephritis, hyperthyroidism and hypothyroidism; Patients with vitiligo or asthma in childhood who have completely relieved and do not need any intervention after adulthood can be included; Asthma requiring medical intervention with bronchodilators cannot be included)
* use of massive dose of glucocorticoids within 4 weeks before enrollment
* laboratory test values do not meet relevant standards within 7 days before enrollment
* significantly lower functions of heart, liver, lung, kidney and bone marrow
* serious or uncontrolled medical diseases or infections
* participating other clinical trial in the same time
* HBsAg (+) and HBV DNA >1×10E3 copiers /mL
* HCV (+) unless HCV RNA PCR(-)
* with any other treatment contraindications

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2022-06-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
3-year progression free survival | 3-year
  time from the randomization to the first disease progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No